CLINICAL TRIAL: NCT03390829
Title: Content and Expectations of Consultations of Patients With Opioid Substitution Treatment Considered as Stabilized: Cross-Testimonials Doctors - Patients (MSOSuiStab)
Acronym: MSOSuiStab
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017-A01752-51
Record Dates: First submitted 2017-10-19; First posted 2018-01-04 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-10

CONDITIONS: Opioid Substitution Treatment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients
  Interventions: Other: semi-directed interviews
- Doctors
  Interventions: Other: semi-directed interviews

INTERVENTIONS:
Other: semi-directed interviews — semi-directed interviews

SUMMARY:
Consultations in general medical practice concerning the follow-up of the patients receiving opiate substitution treatments are not exceptional.

It is nowadays agreed that addictive pathology goes far beyond the issue of product dependence, in favor of a pathology in itself. Centered on problems of attachment, of framework, of trust. The implementation of the opiate substitution treatments and the lifting of the product dependence appears only as a preliminary to the background work with the patient ex-user of opiate.

Finally, the literature provides little information on the experience of general practitioners and their patients under opiate substitution treatments regarding follow-up consultations in the stability phase.

The objective of this work is therefore to study the feelings on follow-up consultations, general practitioners and their patients under opiate substitution treatments considered stabilized.

ELIGIBILITY:
Inclusion Criteria:

* major people patients receiving opiate substitution treatments

Exclusion Criteria:

* considered unstabilized with opiate substitution treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients receiving opiate substitution treatments considered stabilized by their GPs
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-10-20 (Actual); Primary Completion 2019-04-20 (Estimated); Study Completion 2019-04-20 (Estimated)

PRIMARY OUTCOMES:
assessment of feelings on follow-up consultations with standardized questionnaire | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Université Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No